CLINICAL TRIAL: NCT02871843
Title: G-FORCE-1: An Open-Label Phase 1 Two Part Dose Escalation Trial of RRx-001 Concurrent With Radiation and Temozolomide and RRx-001 + Temozolomide Post-RT In Newly Diagnosed Glioblastoma and Anaplastic Gliomas With Intact 1p/19q Chromosomes
Brief Title: RRx-001 + Radiation + Temozolomide In Newly Diagnosed Glioblastoma and Anaplastic Gliomas
Acronym: G-FORCE-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: EpicentRx, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RRx001-17-02
Record Dates: First submitted 2016-08-11; First posted 2016-08-18 (Estimated); Last update posted 2022-05-16 (Actual); Status verified 2022-05

CONDITIONS: Glioblastoma; Oligodendroglioma; Anaplastic Oligodendroglioma
MeSH Terms: conditions — Glioblastoma; Oligodendroglioma | interventions — Temozolomide; Radiation

STUDY DESIGN:
Intervention Model Description: 3+3 Dose Escalation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Escalation of RRx-001 with TMZ + RT (Experimental): Dose escalation of RRx-001 with fixed doses of Temozolomide and radiation followed by Temozolomide maintenance therapy
  Interventions: Drug: RRx-001 dose escalation with TMZ + RT; Radiation: Radiation; Drug: Fixed dose Temozolomide (75 mg/m2); Drug: TMZ Maintenance

INTERVENTIONS:
Drug: RRx-001 dose escalation with TMZ + RT — Dose escalation of RRx-001. Dose levels of 0.5, 1.0, 2.0 and 4.0 mg, once weekly.
Radiation: Radiation — Conformal or intensity-modulated radiotherapy (60 Gy in 2 Gy fractions) given 5 days a week for 30 fractions (about 6 weeks)
Drug: Fixed dose Temozolomide (75 mg/m2) — Oral temozolomide 75 mg/m2 daily for 6 weeks
  Other Names: TMZ
Drug: TMZ Maintenance — TMZ maintenance at 150-200 mg/m2

SUMMARY:
This is a two-part Phase I add-on clinical trial in newly diagnosed glioblastoma or GBM. By "add-on" what is meant is that the experimental intravenous therapy, RRx-001, is combined or "added on" to standard of care. In newly diagnosed GBM standard of care consists of radiotherapy + temozolomide (TMZ) for 6 weeks followed (after a 4-6 weeks break) by maintenance TMZ given until the tumor progresses or worsens. By "maintenance" therapy what is meant is that TMZ is given less frequently to prolong or extend the time during which the tumor remains stable.

G-FORCE-1 will be conducted in two parts; in the first part of the study (Dose Escalation, Part A) patients will be entered or assigned sequentially (that is consecutively) to gradually escalating or increasing doses of RRx-001 after patients have been entered on the previous dose until such time as it is no longer tolerated. At each dose level, a separate cohort or small group of at least 3 evaluable patients will be treated. RRx-001 will be administered by intravenous infusion (in other words, by slow injection in the veins) over 30-45 minutes once weekly during radiotherapy for 6 weeks followed by the FDA-approved chemotherapy, temozolomide (TMZ) alone for up to 6 months or longer.

In the second part of this study (Part B), new groups or cohorts of patients will receive RRx-001 at the dose established in Part A by intravenous infusion over 30-45 minutes once weekly during radiotherapy for 6 weeks. Then, after a 4-6 weeks break, each cohort will receive increasing doses of RRx-001 and temozolomide (in other words, a double dose escalation) to establish an acceptable safety and activity window, in other words, a dose range that is relatively free of toxicity as well as active against the tumor, although the primary purpose of this study is to assess or evaluate safety.

The reason or rationale to "add on" RRx-001 to radiotherapy and TMZ, which is described in more detail below on this page, is as follows: RRx-001 is a radiosensitizer and a chemosensitizer, which means that experimentally it increases the activity of radiation and chemotherapy in tumors. In addition, in other ongoing clinical trials, patients have experienced minimal toxicity or side effects with RRx-001 alone and also in combination with radiation in the brain; therefore, the hope is that RRx-001 will synergize or combine well with radiotherapy and TMZ in GBM without adding toxicity

DETAILED DESCRIPTION:
Glioblastoma multiforme also known by the feared three letter acronym or abbreviation, GBM, is the most common, aggressive and deadly type of brain tumor, which is standardly treated with a combination of radiation and temozolomide (TMZ), an FDA approved chemotherapy agent, followed by temozolomide alone. One of the reasons why glioblastoma is so aggressive and deadly has to do with poor blood flow: it turns out that GBM has multiple inefficient and leaky blood vessels, which leads to ineffective and irregular delivery of nutrients and oxygen to the tumor.

As illogical as it may sound at first, depriving cancer cells of the oxygen and vital nutrients that they need to grow actually makes them more (not less as might be expected) aggressive and harder to treat.

Here's why: for radiation to have an effect on the tumor oxygen is required since the combination of oxygen and radiation produces unstable and highly reactive free radicals; these microscopic free radicals are the equivalent of a spray of bullets, which ricochet or bounce around violently inside the tumor producing catastrophic damage.

Likewise, for chemotherapy such as TMZ to work it has to reach the tumor and when blood vessels are so abnormal that the blood practically ceases to flow the TMZ, for example, may either never actually get there or may arrive in such small quantities that it is ineffective.

The expression "survival of the fittest" also applies: under the poorly oxygenated harsh conditions, which result from this sluggish blood flow only the toughest and most resistant cancer cells survive, making the tumor that much harder to eliminate with traditional therapies.

Think of the blood flow to the tumor as a swamp or a marsh where the rotten water seeps and pools rather than flows and where only the hardiest organisms can compete for scarce resources and low oxygen, which partly explains why this GBM tumor type in particular is often so hard to treat.

This clinical trial, called G-FORCE-1, tests the safety, tolerability and activity of RRx-001, an experimental anticancer agent, with standard radiation and temozolomide followed by temozolomide + RRx-001 in newly diagnosed GBM. Evidence in animals and in human patients with brain metastases, that is cancer cells, which have metastasized or spread to the brain from different locations in the body, has shown that RRx-001, which has many anticancer mechanisms and is generally very well tolerated both alone and in combination with radiation in other clinical trials, increases blood flow to tumors.

The increased blood flow has three possible beneficial consequences: 1) more oxygen is delivered to the tumor, which has the potential to increase the activity of radiation 2) more TMZ makes it to the tumor, which has the potential to increase the activity of TMZ and 3) as conditions in the tumor gradually improve from intolerable or barely tolerable to more acceptable, treatment sensitive cancer cells may start to reappear.

RRx-001 is also thought to work by stimulating the immune system to attack the tumor; tumor biopsies or samples from patients in other RRx-001 trials have demonstrated the infiltration or penetration of a particular kind of white cell called T-cells. As a fourth potentially beneficial consequence of the increased blood flow from RRx-001, these immune T-cells may have better access to the tumor, which may, in turn, increase killing of the cancer cells.

G-FORCE-1 is a Phase 1 trial, which means that the main endpoint is to test the safety and tolerability of RRx-001 in combination with radiation and temozolomide and not its activity; however patients will be followed for responses to treatment and overall survival

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven diagnosis of high-grade glioma, including anaplastic glioma (WHO grade III with 1p/19q chromosomes intact), glioblastoma (WHO grade IV) or gliosarcoma (WHO Grade IV);
* The tumor must not have an infratentorial component;
* The patient must have recovered from the effects of surgery, postoperative infection and other complications before enrollment;
* Estimated survival of at least 12 weeks;
* Karnofsky Performance Score of ≥ 70% at the time of entry
* Stable or decreasing steroid dose within 2 weeks of first dose of study drug if patient is taking steroids. No steroid use is also acceptable.
* Neurological stability for at least 14 days prior to first dose of study drug;
* Acceptable liver function at Screening,
* Serum creatinine < 1.5x institution upper limit of normal
* Acceptable hematologic status at Screening
* Female subjects of childbearing potential, and male subjects with partners of childbearing potential, must agree to use medically acceptable methods of contraception.

Exclusion Criteria:

* Prior invasive malignancy (except for non-melanomatous skin cancer) unless disease free for ≥ 3 years.
* Recurrent malignant gliomas previously treated with radiotherapy and/or chemotherapy
* Metastases detected below the tentorium or beyond the cranial vault, including tumors with evidence of leptomeningeal metastases as previously indicated;
* Prior chemotherapy or radiosensitizers for cancers of the head and neck region; note that prior chemotherapy for a different cancer is allowable, except prior temozolomide. Prior use of Gliadel wafers or any other intratumoral or intracavitary treatment are not permitted;
* Prior radiotherapy to the head or neck (except for T1 glottic cancer), that would result in overlap of radiation fields.
* Active connective tissue disorders, such as lupus or scleroderma that in the opinion of the treating physician may put the patient at high risk for radiation toxicity;
* Unresolved toxicity higher than CTCAE (v. 4.03) Grade 1 attributed to any prior therapy/procedure excluding alopecia and hypothyroidism;
* Acquired immune deficiency syndrome (AIDS) due to the potential for increased complications from treatment; note, however, that HIV testing is not required
* No other concurrent chemotherapeutic or investigational agents for this cancer. However, concurrent glucocorticoids are allowed;
* Inability to swallow pills;
* Serious co-morbid medical conditions, or a clinically significant laboratory finding(s) or any finding(s) on history and/or examination that, in the opinion of the Investigator, could interfere with the conduct of the study or could put the patient at unacceptable risk;
* Patients who are pregnant or lactating or who are planning to become pregnant during the course of the study are excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2017-02-14 (Actual); Primary Completion 2019-10-11 (Actual); Study Completion 2021-09-19 (Actual)

PRIMARY OUTCOMES:
Number, frequency and type of adverse events | 12 weeks

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | 4 months
  Objective Response rate as determined by the patient's best tumor response, Duration Of Response (DOR) and Time To Progression (TTP) using modified RANO criteria
Clinical Benefit Rate (CBR) | 4 months
  Clinical Benefit Rate as determined by the patient's best tumor response, Duration Of Response (DOR) and Time To Progression (TTP) using modified RANO criteria
Intracranial Progression Free Survival | 4 months
  Intracranial PFS is defined as the time that a patient lives with intracranial tumors before progression. Changes in intracranial tumors will be measured by MRI and scored using RANO criteria. The response assessment will take into account MacDonald Criteria using bi-dimensional measurements of the largest contrast- enhancing area, RANO Criteria, FLAIR imaging and clinical status.
Overall Survival | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Bryan Oronsky, Study Director — Chief Medical Officer
Locations (3):
- United States (3):
  - University of California San Francisco (UCSF), San Francisco, California
  - The Cancer Institute of New Jersey (Rutgers University), New Brunswick, New Jersey
  - Weill Cornell Brain Tumor Center, New York, New York